CLINICAL TRIAL: NCT00002135
Title: An Open-Label Safety Study of Oral Ganciclovir Maintenance Treatment of CMV Retinitis in People With Limited Venous Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 037C; GANS2224
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-11

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Ganciclovir; Administration, Oral; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To provide oral ganciclovir to patients who require maintenance for control of cytomegalovirus (CMV) retinitis, but who lack patent permanent central venous access for long-term administration of intravenous drugs.

DETAILED DESCRIPTION:
Patients receive oral ganciclovir as maintenance. Patients enrolled at time of closure of enrollment will receive 2 months of study drug and undergo follow-up.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS.
* Stable CMV retinitis.
* Treatment with IV ganciclovir or IV foscarnet for at least 18 of the past 21 days.
* No permanent central IV catheter at present.
* Had a permanent central IV catheter removed two or more times within the past 6 months due to catheter infection or thrombosis.
* Consent of guardian if less than legal age of consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Require continuation of concomitant medications precluded by this protocol.

Concurrent Medication:

Excluded:

* Intravitreal anti-CMV treatment.
* Any other concomitant medications precluded by the protocol.

Patients with the following prior condition are excluded:

History of hypersensitivity to acyclovir or ganciclovir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Roche Global Development - Palo Alto, Palo Alto, California, United States

REFERENCES:
- [Background] Intravenous versus oral ganciclovir: European/Australian comparative study of efficacy and safety in the prevention of cytomegalovirus retinitis recurrence in patients with AIDS. The Oral Ganciclovir European and Australian Cooperative Study Group. AIDS. 1995 May;9(5):471-7. PMID 7639972
- [Background] Drew WL, Ives D, Lalezari JP, Crumpacker C, Follansbee SE, Spector SA, Benson CA, Friedberg DN, Hubbard L, Stempien MJ, et al. Oral ganciclovir as maintenance treatment for cytomegalovirus retinitis in patients with AIDS. Syntex Cooperative Oral Ganciclovir Study Group. N Engl J Med. 1995 Sep 7;333(10):615-20. doi: 10.1056/NEJM199509073331002. PMID 7637721